CLINICAL TRIAL: NCT06807957
Title: Effectiveness of Inspiratory Muscle Training on Respiratory Muscle Strength and Physical Performance in Amateur CrossFit® Athletes: A Randomized Controlled Trial
Brief Title: Inspiratory Muscle Training in Amateur CrossFit® Athletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of the Valleys of Jequitinhonha and Mucuri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 81443024.9.0000.5108
Record Dates: First submitted 2025-01-17; First posted 2025-02-04 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: Sport; Athlete; Respiratory muscles; CrossFit

STUDY DESIGN:
Intervention Model Description: The randomization sequence for the experimental and control groups, with a 1:1 allocation ratio, will be generated by computer software by one of the researchers who will not be involved in participant recruitment. The groups will be coded, and the allocation will be transferred to a series of sequentially numbered, sealed, opaque envelopes.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with IMT (Experimental): CrossFit® Training: ParticipaIMT: The intervention will utilize the POWERbreathe® device. Participants will be provided with the device for home training. The model selected for this study is the POWERbreathe® Classic Medium Resistance (Fitness).
  The load will be set at 50% of each participant's MIP, as determined during the assessment phase using a vacuum manometer. IMT will be performed in two sets of 30 breaths through a mouthpiece connected to the POWERbreathe®, with a one-minute rest between sets. Participants will complete the training five days per week at home over the course of eight weeks. Additionally, participants will monitor their adherence by completing a log sheet to mark training days. To ensure proper use and management of the device, each participant will receive individual training after randomization. At the end of the eight weeks, participants will return the equipment to the research team for cleaning and redistribution to another participant in the same group.
  Interventions: Device: Group with IMT; Behavioral: CrossFit® Training
- Group without IMT (Placebo Comparator): Group without IMT Participants allocated to the "No IMT Group" will receive the same interventions as the "IMT Group," except for respiratory training. These participants will continue attending CrossFit® training sessions at the gym. They will also perform a simulated IMT, using a device without the valve that generates resistance to the respiratory muscles.
  Interventions: Behavioral: CrossFit® Training

INTERVENTIONS:
Device: Group with IMT — Group with IMT + CrossFit training
  Arms: Group with IMT
Behavioral: CrossFit® Training — The training routine will occur seven days a week, with participants encouraged and motivated to attend at least five training sessions. CrossFit® classes will include: warm-up exercises, strength training (with a focus on Olympic weightlifting and free weights), strength endurance (body weight and external loads), aerobic capacity (across multiple domains), maximal aerobic power (across multiple domains), anaerobic capacity (across multiple domains), cool-down activities, and mobility exercises. Each training session will be designed and supervised by a team of certified physical educators.

SUMMARY:
The aim of this randomized controlled trial is to investigate the effectiveness of inspiratory muscle training (IMT) on the performance of athletes in CrossFit® activities, respiratory muscle strength, and perceived post-training fatigue. This study follows a two-arm randomized controlled trial protocol. Ninety-four volunteers aged between 18 and 60 years, enrolled in CrossFit® training, will be randomly allocated to the IMT Group, which involves respiratory training using a linear load device (Powerbreathe®) in conjunction with CrossFit® training; or the Non-IMT Group, which undergoes the same training as the intervention group but uses a device without a valve that ensures resistance. The primary outcome is to investigate the effectiveness of IMT: on maximum inspiratory pressure and maximum expiratory pressure. The secondary outcomes include performance in the six-minute walk test, Pistol, Burpee, Sit-up, Box Jump, Thruster, and Single-Under, burning 25 calories on the "Air Bike" measured by the time taken to reach the 25-calorie mark on this equipment, as well as the assessment of subjective fatigue perception. All outcomes of interest will be collected at baseline and reassessed: mid-term (8 weeks after allocation); and long-term (12 weeks after allocation), the IMT and MEP will be reassessed. Analyses will follow the intention-to-treat principle. Treatment effects will be assessed using Linear Mixed Models. The results of this study may help clarify the effects of IMT on CrossFit® athletes.

DETAILED DESCRIPTION:
Study design: This is a prospective randomized controlled trial with two arms. The study was registered with the Research Ethics Committee of the Universidade Federal dos Vales do Jequitinhonha e Mucuri (UFVJM): 81443024.9.0000.5108. Procedures and data collection: Participants who seek the CrossFit® service and enroll, as well as those who are already enrolled, will be invited to participate in this study. All eligible participants will receive information about the study and must sign an informed consent form before participating. The initial assessment and reassessment of the participant will take place at Academia Compasso Sete Lagoas (Boa Vista Unit and/or Centro Unit). The data collected will be: age, height, weight, body mass (BM), Body Mass Index (BMI), heart rate, blood pressure, gender, smoking history (yes/no), medications in use, time practicing the sport and the presence of any comorbidities. All outcomes of interest (respiratory muscle strength, subjective perception of fatigue and results obtained in CrossFit® exercises) will be collected at baseline and reassessed at the following time points: medium term (8 weeks after allocation) and long term (12 weeks after allocation), in an assessment room at the gym. The collected data will initially be entered into a standardized data collection form and then transferred to an Excel table.

The evaluation process will be divided as follows: first, the participant will complete the evaluation form, and then their MIP and MEP values will be collected. Next, the first evaluation test will be performed: "Air Bike" (25 calories); then the evaluation sequence will be performed: Sit-up, Pistol, Burpee, Box Jump, 6MWT, Thruster, and Single-Under. Additionally, after completing all the exercises on the second day of evaluation, the Borg Scale will be administered.

The randomization sequence for the experimental and control groups, with an allocation ratio of 1:1, will be generated by a computer program by one of the researchers who will not be involved in the recruitment of participants. The groups will be coded and the allocation will be transferred to a series of sealed and sequentially numbered opaque envelopes. Two evaluators participated in this stage of the research: researcher 1 will be responsible for the evaluations; and researcher 2 for randomization and distribution of equipment.

Group with TMI: CrossFit® training: participants will be guided and encouraged to attend at least 5 days of training. TMI: the device used for the intervention will be the POWERbreathe®. The load used will be 50% of MIP. The TMI will be performed in two series of 30 breaths through the mouth through the mouthpiece connected to the POWERbreathe®, with a 1-minute interval between series.

Group without TMI: participants allocated to the "No TMI Group" will receive the same interventions as the "Group with TMI", but without the respiratory training included. In addition, they will also perform the TMI in a simulated manner.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years;
* Be enrolled in a CrossFit® program;
* Be available to perform TMI at home 5 days a week.

Exclusion Criteria:

* Have any musculoskeletal, cardiovascular and/or neurological condition that prevents CrossFit® and/or IMT from being performed;
* Be a smoker;
* Not sign the Termo de Consentimento Livre Esclarecido (TCLE);
* Be performing or have performed IMT using linear load equipment in the last month.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength (Maximum inspiratory pressure (MIP) | at 8 weeks and 12 weeks
  Respiratory muscle strength (Maximum inspiratory pressure (MIP) Description: The assessment of the strength of the resistant muscles will be performed using a vacuum manometer with an operating range of ± 300 cmH2O. To measure the MIP, the participant must exhale until reaching their Residual Volume (RV), immediately connecting the mouthpiece to the oral tract and making a maximum inspiratory effort against the occluded airway, holding for at least one second.
Respiratory muscle strength (Maximum expiratory pressure (MEP)) | at 8 and 12 weeks
  The assessment of the strength of the resistant muscles will be performed using a manovacuometer with an operating range of ± 300 cmH2O. To measure MEP, the participant must inhale until reaching their Total Lung Capacity and then, inserting the mouthpiece into the oral cavity, perform a maximum expiratory effort against the occluded airway, which must be maintained for at least one second.

SECONDARY OUTCOMES:
Subjective perception of effort | at 8 weeks
  At the end of the exercises on the second day of evaluation, study participants must respond/quantify their perception of effort after training - using the Borg's Perceived Exertion Scale (Scale Borg / 6 - 20). The higher the score, the greater the feeling of effort
6-minute walk test (6MWT) | at 8 weeks
  The 6MWT is a commonly used test for objective assessment of functional exercise capacity. In this relatively low complexity test, the patient is asked to walk as far as possible along a 30 m corridor for a period of 6 minutes, with the primary outcome being the walking distance during the 6 minutes
Box Jump | at 8 weeks
  Standardization of 60 repetitions with timed timing. Height for male population: 60 centimeters (cm); Height for female population: 50 cm
Sit Up | at 8 weeks
  Maximum repetitions in a 2-minute period. In the starting position, the participant will have their back straight and lying on the floor. The hands should be touching the floor behind the head and the legs should be in the "Butterfly" position. The participant should raise the torso, flexing the spine, lifting the shoulders off the floor, until the hands touch the floor with the feet. Then, the upper part of the body should return to the starting position. The participant should perform as many movements as possible within a time of 2 minutes, with the number of repetitions recorded.
Burpee | at 8 weeks
  Maximum repetitions in a 2-minute period. Initially, the participant will be in an upright position, then he/she must perform a squat with his/her hands on the floor. After that, he/she must extend his/her elbows and push his/her legs back, keeping his/her hands in the same place, to get into a plank position. Then, a full push-up must be performed. With another small jump, the participant must return to the position of step 2, with his/her hands and feet on the floor. Finally, use all his/her strength and momentum to perform a vertical jump. The participant must perform as many repetitions as possible in a maximum period of 2 minutes, with the number of repetitions recorded
Pistol | at 8 weeks
  Maximum repetitions in a 2-minute period. The participant must perform as many repetitions of the movement as possible with the right and/or left leg in a maximum of 2 minutes. Standing with arms extended forward, the participant must extend one leg forward. The leg that will remain in support will perform the squat movement, keeping the other leg always extended. The abdomen must remain contracted and the leg extended throughout the squat movement. The torso must lean forward, while the hips are positioned backward. The knee must always be forward, in the direction of the toes. After the squat, return to the starting position.
Single-Under | at 8 weeks
  Standardization of 200 jumps with timed timing.
Thruster | at 8 weeks
  20 repetitions with timed exercise. Men's load: 95lb - 25lb on each side; Women's load: 65lb - 15lb on each side
Effectiveness of TMI on race performance: 25 calorie expenditure on the Air Bike | at 8 weeks
  Before starting the test, the evaluator will adjust the seat to hip height and ensure that each participant's arms can comfortably reach the handles. The participant must then perform synchronous movements of the upper and lower limbs until reaching the 25-calorie mark

CONTACTS AND LOCATIONS:
Locations (1):
- Academia Compasso - Kapura, Sete Lagoas, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the publication of results. These data will be available in the database: Open Science Framework
Supporting Information: Study Protocol
Time Frame: Unending (Starting after publication with no end date)
Access Criteria: Researchers in the area who are interested